CLINICAL TRIAL: NCT05945329
Title: A Prospective, Randomized, Controlled, Multi-Center Study of GalaFLEX LITE™ Scaffold in Treatment of Capsular Contracture After Breast Implant Augmentation
Brief Title: Study of GalaFLEX LITE™ Scaffold in Treatment of Capsular Contracture After Breast Implant Augmentation
Acronym: STANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DVL-BR-001
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Capsular Contracture Associated With Breast Implant; Capsular Contracture Grade III; Capsular Contracture Grade IV

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, randomized
Who Masked: Participant
Masking Description: Participant will not be made aware of whether they receive standard-of-care surgery or surgery with the study device. They will be made aware at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- GalaFlex Light Scaffold (Experimental): Surgery performed with GalaFlex Lite Scaffold.
  Interventions: Device: GalaFLEX LITE™ Scaffold
- Standard Surgery (Active Comparator): Surgery performed using standard surgical procedures with no scaffold.
  Interventions: Other: Standard surgery

INTERVENTIONS:
Device: GalaFLEX LITE™ Scaffold — Bioabsorbable surgical mesh manufactured from poly-4-hydroxybutyrate (P4HB) and knitted into a surgical scaffold used to reinforce soft tissue
  Arms: GalaFlex Light Scaffold
Other: Standard surgery — Surgery performed without the use of a scaffold
  Arms: Standard Surgery

SUMMARY:
Prospective, randomized, controlled study to assess the safety and effectiveness of GalaFLEX LITE™ Scaffold in revision surgery for reduction of capsular contracture recurrence and/or malposition in implant-based breast augmentation patients versus patients undergoing conventional revision surgery with no supportive matrix or acellular dermal matrix (ADM). Subjects will be randomized 2:1 to receive either GalaFLEX LITE™ Scaffold or standard care (no ADM or matrix placement). This study is designed using an adaptive approach. The number of the treated breasts will range between 250 and 530.

DETAILED DESCRIPTION:
Capsular contracture is the number one complication leading to revision surgery after breast augmentation(2-4) which has been commonly cited as impacting 10 to 20% of all breast augmentation patients.(5-10) A prospective, randomized controlled study of patients presenting with Baker grade III or IV capsular contracture will be undertaken to investigate the ability of P4HB (specifically GalaFLEX LITE™ Scaffold) to reduce the recurrence of clinically significant CC and/or malposition requiring surgical correction. The primary endpoint is a composite of capsular contracture recurrence and/or breast implant malposition recommended for surgery OR breast infections requiring oral or IV antibiotic treatment within 90 days of surgery and/or peri-implant fluid collection needing a drainage procedure within 10-90 days of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Genetically female ≥22 and ≤66 years of age;
2. Breast augmentation subject with capsular contracture (Baker grade III or IV);
3. Desired a new implant with no more than a 25% increase in implant size (not to exceed a volume increase greater than 150cc compared to the existing implant);
4. Planned revision approach via inframammary fold (IMF) incision;
5. Willing and able to comply with the study procedures including the 2-year follow-up visit;
6. Lives within 3 hours driving distance from the investigator site; and,
7. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. BMI <18 or >35
2. Existing and/or replacement implant size > 800 cc
3. Had ≥2 capsular contracture revisions on the breast(s) intended for treatment
4. Has an extra-capsular rupture (breast implant silicone gel or saline has leaked outside of the capsule) in breast(s) intended for treatment
5. Has prior use of a matrix (synthetic or biologic) in the breast(s) intended for treatment.
6. Abnormal findings on diagnostic imaging within 1-year of study enrollment (mammogram for patients ≥35 years old; MRI for patients <35 years old or breast ultrasound if MRI is contraindicated)
7. Has symptoms consistent with Breast Implant Illness (BII)Systemic Symptoms Associated with Breast Implants (SSBI)
8. Infection present in the breast (day of surgery exclusions are noted in Section 5.3)
9. Current or recent breast feeding (within 3-months or enrollment) or history of mastitis within the 6-months prior to enrollment
10. Prior or current diagnosis of breast cancer
11. Has a mass that was palpated and has not been determined benign via acceptable imaging (MRI) or biopsy results
12. Has undergone prior chest radiation treatment
13. Has received chemotherapy within the last 12 months
14. Current or recent (within 1-year of enrollment) alcohol/substance abuse
15. Current or recent (within 4-weeks of enrollment) nicotine user (includes cigarettes, vaping, patches, gum, etc.)
16. History of Breast Implant-Associated Anaplastic Large Cell Lymphoma (BIA-ALCL) or Breast Implant Associated Squamous Cell Carcinoma (BIA-SCC)
17. Planned use of another type of matrix (such as ADM) in addition to GalaFLEX LITE™
18. Current or planned use of medical (e.g. Singulair), physical (e.g. massage), or device-assisted (e.g. mechanical/thermal ultrasound) tools to manage the breast capsule(s)
19. Any medical condition that, in the opinion of the investigator, may be associated with unduly high risk of intra- or post-operative complications (e.g., insulin-dependent diabetes, autoimmune disease, connective tissue disorder, chronic lung or severe cardiovascular disease)
20. Concurrent or planned (within the 2-year follow-up time period) elective cosmetic breast operation to the treated breast (e.g., autologous fat transfer, mastopexy, or implant size changes)
21. Currently enrolled or has plans to enroll in another clinical study that would interfere with this study, unless it is a retrospective or observational study
22. Is pregnant or plans to become pregnant during the study period
23. Known allergy to tetracycline hydrochloride and kanamycin sulfate
24. Any condition that, in the Investigator's opinion, would preclude the use of the study device, interfere with the evaluation of the device or breast related outcomes
25. Subject will not remain under the care of the investigator for all plastic surgery procedures while enrolled in the study
26. Actively using immunosuppressants such as oral steroids or biological therapies (inhalers or topical steroids are permitted)
27. Confirmed diagnosis of the following rheumatic diseases or syndromes: systemic lupus erythematosus, Sjorgren's syndrome, scleroderma, polymyositis, or any connective tissue disorder, rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondyloarthropathies, any other inflammatory arthritis, fibromyalgia, or chronic fatigue syndrome
28. Has, in the investigator's opinion, a mental illness or disability that would preclude their participation in the study
29. Subject has an implant that was never commercially available in the United States (had their breast augmentation in another country)
30. Has been implanted with any silicone implant other than breast implants
31. Is taking any drugs that would interfere with blood clotting or might result in elevated risk of significant postoperative complications
32. Works for Sponsor or any of their subsidiaries, the study surgeon, or is helping to conduct the study or are directly related to anyone that works for BD or any of their subsidiaries or the study surgeons. -

Ages: 22 Years to 66 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Genetically female
Enrollment: 250 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of GalaFLEX LITE™ Scaffold for the stabilization of the implant pocket | 24-months after index surgery
  Composite of Recurrent Capsular Contracture Baker grade III/IV and/or breast implant malposition

SECONDARY OUTCOMES:
Patient quality of life and satisfaction (12-month) | 12-months after index surgery
  Select Breast-Q© modules (standardized patient survey) for the treated breast(s): psychosocial wellbeing; sexual wellbeing; satisfaction with breasts; and physical wellbeing - chest
Patient quality of life and satisfaction | 24-months after index surgery
  Select Breast-Q© modules (standardized patient survey) for the treated breast(s): psychosocial wellbeing; sexual wellbeing; satisfaction with breasts; and physical wellbeing - chest
Safety of GalaFLEX LITE™ Scaffold for the stabilization of the implant pocket, reduction of capsular contracture recurrence, and/or malposition | 90 days
  The occurrence of:
  * Breast fluid collection requiring a drainage procedure at any time, or after drain removal if one is used, within 90 days of surgery
  * Breast infection requiring oral (PO) or intravenous (IV) antibiotics related to the contracture revision surgery within 90 days of surgery

OTHER OUTCOMES:
Device or procedure related adverse events | 24-months after index surgery
  Select adverse events including: breast infection requiring PO or IV antibiotics related to the revision surgery; breast fluid collection requiring a drainage procedure; breast implant loss; any unscheduled/unanticipated breast reoperation; breast implant malposition recommended for surgery; skin necrosis; wound dehiscence; any seroma within 90 days of surgery; any hematoma within 90 days of surgery; capsular contracture Baker Grade >1; and red breast syndrome

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Defyne MD, Scottsdale, Arizona
  - The Practice Plastic Surgery, Beverly Hills, California
  - California Aesthetic Center, Huntington Beach, California
  - Donald S Mowlds, MD A Professional Corporation, Newport Beach, California
  - Newport Plastic and Reconstructive Surgery Associates, Newport Beach, California
  - Stewart Wang MD Inc., Pasadena, California
  - Tim Sayed MD, San Diego, California
  - Sanctuary Plastic Surgery, Boca Raton, Florida
  - Careaga Plastic Surgery, Miami, Florida
  - Aesthetic Enhancements Plastic Surgery, Orlando, Florida
  - Billington Plastic Surgery, St. Petersburg, Florida
  - VIVIFY Plastic Surgery, Tampa, Florida
  - The Graivier Center, Alpharetta, Georgia
  - Monarch Plastic Surgery and Skin Renewal Center, Atlanta, Georgia
  - Meridian Plastic Surgery Center, Indianapolis, Indiana
  - Reno Tahoe Plastic Surgery, Reno, Nevada
  - VIP Plastic Surgery, West Long Branch, New Jersey
  - Plastic Surgery Institute of New York, New York, New York
  - H/K/B Surgery, Huntersville, North Carolina
  - Essential Medical Research, Tulsa, Oklahoma
  - Pittsburgh Center for Plastic Surgery, Pittsburgh, Pennsylvania
  - The Plastic Surgery Center of Nashville With HKB, Nashville, Tennessee
  - Farah Naz Khan, Dallas, Texas
  - Southwest Plastic Surgery, El Paso, Texas
  - Aesthetic Center for Plastic Surgery, Houston, Texas
  - Hill Country Plastic Surgery, San Antonio, Texas
  - Next Stage Clinical Research, San Antonio, Texas
  - The Plastics Clinic, Draper, Utah
  - Athenix Advanced Plastic Surgery & Aesthetic Center, Seattle, Washington
  - Allen Gabriel MD, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No